CLINICAL TRIAL: NCT03475979
Title: Surveillance for Second Breast Cancer With Abbreviated Breast MRI, Ultrasound, and Mammography in Women With BRCA Mutation Testing
Brief Title: Abbreviated Breast MRI for Second Breast Cancer Detection in Women With BRCA Mutation Testing
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Korean Society of Breast Imaging & Korean Society For Breast Screening (Unknown); Bayer (Industry)
Responsible Party: Principal Investigator, Woo Kyung Moon, Professor, Seoul National University Hospital
Other Study IDs: AB-MR for Second Breast Cancer
Record Dates: First submitted 2018-03-13; First posted 2018-03-23 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Breast Cancer; BRCA1 Mutation; BRCA2 Mutation; Recurrent Breast Cancer; Metachronous Neoplasm
MeSH Terms: conditions — Breast Neoplasms; Neoplasms, Second Primary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study Purpose:

A multicenter prospective study to evaluate the outcome of second breast cancer surveillance with abbreviated breast MR (AB-MR) or ultrasound (US) in addition to annual mammography in women with BRCA1/2 mutation testing

Study Scheme:

* AB-MR, US, and digital mammography will be performed on the same day and interpreted independently at baseline and then after 1 year.
* After completion of study, patients are followed-up for at least 1 year.

DETAILED DESCRIPTION:
For women with a BRCA1/2 mutation who are treated for breast cancer, screening of remaining breast tissue with annual mammography and breast MRI is recommended. For women who met BRCA testing criteria but show an uninformative negative result or a variant of unknown significance (VUS) result, there is no established recommendation for second breast cancer surveillance.

Abbreviated breast MRI (AB-MR) is a fast and low-cost examination that show equivalent diagnostic accuracy to that of the standardized dynamic protocol breast MRI. Breast ultrasound (US) can detect additional cancers that are occult on mammography and is indicated in high-risk patients who cannot tolerate MRI.

The purpose of this multicenter prospective study is to evaluate the outcome of second breast cancer surveillance with AB-MR or US in addition to annual mammography in women with BRCA1/2 mutation testing.

AB-MR, US, and digital mammography will be performed on the same day at baseline and then after 1 year and images will be interpreted independently according to the Breast Imaging Reporting and Data System (BI-RADS) by experienced radiologists. The BI-RADS category 3 or higher is defined as test-positive. The reference standard will be a biopsy or at least 1 year of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 25 years and 75 years with a personal history of breast cancer
* BRCA mutation test done (meeting any of the following criteria): 1) early-age-onset breast cancer (40 years or younger), 2) bilateral breast cancers (synchronous) 3) personal history of ovarian cancer and/or other multiple primary cancers 4) family history of breast and/or ovarian cancer in first- or second-degree relatives
* No symptom or sign of secondary breast cancer (no palpable mass, bloody nipple discharge, abnormal skin change, nipple retraction)
* Written informed consent is given

Exclusion criteria:

* Initial breast cancer stage IV
* Bilateral mastectomy done
* Diagnosis of second breast cancer or regional/distant metastasis
* Systemic chemotherapy for any cancer
* Pregnant or lactating
* Contraindication to breast MRI with contrast enhancement

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients who met BRCA testing criteria and undergo post-operative surveillance for secondary breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 1564 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity (co-primary) | 1 year
  To compare the sensitivity and specificity of AB-MR, US, and mammography for the detection of secondary breast cancer

SECONDARY OUTCOMES:
Cancer detection rate (CDR) | 1 year
  To compare the CDR (no. of detected cancers/1,000 examinations) of AB-MR, US, and mammography
Positive predictive value (PPV) | 1 year
  To compare the PPV (no. of detected cancers / no. of positive examinations) of AB-MR, US, and mammography
Negative predictive value (NPV) | 1 year
  To compare the NPV (no. of detected cancers / no. of negative examinations) of AB-MR, US, and mammography
Histopathologic characteristics of secondary breast cancers | 1 year
  To describe the histologic type, tumor grade, and molecular tumor subtype of secondary breast cancers detected at AB-MR, US, and mammography

CONTACTS AND LOCATIONS:
Overall Officials: Woo Kyung Moon, MD, PhD, Principal Investigator — Professor
Locations (1):
- Seoul National University Hospital, Seoul, South Korea